CLINICAL TRIAL: NCT00843388
Title: A Randomized Doubleblind Placebo Controlled Crossover Study With Hexalacton in Patients With Type 1 Diabetes and Microalbuminuria
Brief Title: A Crossover Study With Hexalacton in Patients With Type 1 Diabetes and Microalbuminuria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Peter Rossing, Steno Diabetes Center, Dep 520
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2306; Eudra CT: 2008-004839-38
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes Mellitus; Nephropathy; Blood Pressure
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 60 days treatment with tablet hexalacton 25 mg OD.
  Interventions: Drug: Spironolacton (hexalacton(R))
- 2 (Placebo Comparator): Inactive drug of 25 mg OD
  Interventions: Drug: placebo tablet

INTERVENTIONS:
Drug: Spironolacton (hexalacton(R)) — Tablet Spironolacton 25 mg OD
  Arms: 1
Drug: placebo tablet — placebo tablet 25 mg OD
  Arms: 2

SUMMARY:
A double blind, randomized, cross over study in type 1 diabetic patients. 20 patients, age 18-65 years is treated with spironolacton (Hexalacton (R)) for 60 days followed by 60 days treatment with placebo(or opposite). Primary aim: albuminuria, an expected decrease during hexalacton treatment. Secondary aim: ambulatory blood pressure, GFR, plasma-renin, angiotensin, aldosteron.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* age 18-80 years
* microalbuminuria

Exclusion Criteria:

* blood pressure> 160/100 mmHg
* persistent macroalbuminuria
* pregnancy or in risc of this
* P-Potassium>5.7 mmol/l
* Eplerone treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
albuminuria, expected decrease | 60 days

SECONDARY OUTCOMES:
GFR | 60 days
ambulatory blood pressure | 60 days
plasma renin, angiotensin, aldosteron | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: stine e nielsen, MD, Principal Investigator — Steno Diabetes Center Copenhagen